CLINICAL TRIAL: NCT03251599
Title: The Effect of Two Different Rates of Nitroglycerin Infusion on Cerebral Rewarming During Rewarming Period of Hypothermic Cardiopulmonary Bypass
Brief Title: The Effect of Nitroglycerin Infusion Rate on Cerebral Rewarming During Hypothermic Coronary Artery Bypass Grafting
Acronym: nitrotherm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Asst. Prof. of Anesthesiology and Reanimation, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017/5
Record Dates: First submitted 2017-08-01; First posted 2017-08-16 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Bypass; Cardiopulmonary Bypass
Keywords: peak temperature; rewarming rate; surgical outcomes
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: Intervention type is drug dosage. Patients will be assigned to 2 arms, where they will receive different doses of the same drug. The study will end when both of the arms will have at least 48 patients each.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be via enclosed envelope technique. The anesthetic management of the patient will be provided by an anesthesiologist other than the investigator. This anesthesiologist will not be blinded to the dose of the study drug, and will be responsible from the administration of the appropriate dose of the study drug.
  The perfusionist, who is the main care provider during the rewarming period of the cardiopulmonary bypass, will be blinded to the dose of the study drug.
  The investigator will be blinded, and will be responsible from the collection, and validation of the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glyceryl trinitrate 0.2 (Sham Comparator): Drug Intervention Generic name: Glyceryl trinitrate Dosage form: Ampoule for intravenous infusion Dosage: 0.2 mcg/kg/minute Frequency and duration: The infusion will start as soon as the rewarming period starts, will continue throughout the operation and throughout the first 24 hours of the postoperative period.
  Interventions: Drug: Glyceryl trinitrate 0.2
- Glyceryl trinitrate 0.5 (Active Comparator): Drug Intervention Generic name: Glyceryl trinitrate Dosage form: Ampoule for intravenous infusion Dosage: 0.5 mcg/kg/minute Frequency and duration: The infusion will start as soon as the rewarming period starts, will continue throughout the operation and throughout the first 24 hours of the postoperative period.
  Interventions: Drug: Glyceryl trinitrate 0.5

INTERVENTIONS:
Drug: Glyceryl trinitrate 0.2 — These patients will receive glyceryl trinitrate infusion at a rate of 0.2 mcg/kg/min throughout the rewarming period of cardiopulmonary bypass, which usually lasts for 30-45 minutes.
  Other Names: Nitroglycerin, Perlinganit
  Arms: Glyceryl trinitrate 0.2
Drug: Glyceryl trinitrate 0.5 — These patients will receive glyceryl trinitrate infusion at a rate of 0.5 mcg/kg/min throughout the rewarming period of cardiopulmonary bypass, which usually lasts for 30-45 minutes.
  Other Names: Nitroglycerin, Perlinganit
  Arms: Glyceryl trinitrate 0.5

SUMMARY:
Glyceryl trinitrate is used in coronary artery bypass grafting surgery. This surgery frequently employs hypothermic cardiopulmonary bypass, where the whole body is cooled down to 28-32 °C to arrest the heart, and protect the organs from ischemic insult. When the cardiac repair or grafting is done, the body is warmed to 37 °C. During this "rewarming period", the heart has to beat against the vessels, all of which are constricted due to hypothermia.

To overcome this constriction of the vessels, and decrease the workload of the heart, glyceryl trinitrate is infused. This drug causes significant dilatation in arteries and veins, which allows the heart to pump the blood with less force. The dilatation of the vessels also allows the body to rewarm more easily.

The investigators' concern is whether increased infusion rates of glyceryl trinitrate may cause uncontrolled rewarming of the brain or not. The investigators will measure the temperature of the brain using a temperature probe located in the nasal cavity. The temperature will be recorded at each minute during the the rewarming period. Results of two commonly used infusion rates of glyceryl trinitrate will be compared.

DETAILED DESCRIPTION:
Hypothermia had demonstrated potential benefits in myocardial infarction, organ transplantation, and cardiopulmonary bypass. The brain uses 2/3 of the oxygen it receives to support cerebral electrophysiological function, while the rest is used for maintenance of cellular integrity. Anesthetic drugs alter only the first portion, while temperature is the only agent known to affect both portions (the cerebral consumption of oxygen decreases 6-7 % per degree centigrade reduction in temperature).

Although hypothermia is effectively used to protect the brain and myocardium from ischemia, studies report that rapid rewarming is correlated with brain injury. Therefore it is common practice to monitor the nasopharyngeal temperature and to keep the gradient between heat-exchanger and nasopharynx during rewarming at 2-3 °C.

This study's main concern is that the infusion rate of glyceryl trinitrate may affect the rewarming rate of the body and the brain during te rewarming period. One possibility is that the increased vasodilatation resulting from glyceryl trinitrate may divert most of the heat to the body and protect the brain from overheating. The other possibility is that the increased partial pressures of carbon dioxide may render the brain more susceptible to the vasodilatatory actions of glyceryl trinitrate, which may cause the brain to overheat.

This study will measure temperatures at several sites of the patient and the cardiopulmonary bypass machine:

* Nasopharynx: a probe inside the nasal cavity, located above the palate.
* Core temperature: a probe inside the esophagus, 12 cm distal from where the heart and breath sounds are heard best.
* Heat-exchanger: recorded as is supplied by the heat exchanger as the temperature of the water inside the heat exchanger.
* Returning blood: measured at the entrance of reservoir
* Blood leaving the oxygenator: measured at the outlet of the oxygenator

All patients scheduled for cardiopulmonary bypass grafting surgery, and aortic arch surgery will be recruited.

Data will be collected by an observer blinded to the glyceryl trinitrate dose used. Data management will be done via an electronic database including demographic data, anesthetic records, and bypass records of the patient. All data will be anonymized on a case-by-case fashion after the surgery. Data analysis will be performed using R statistical software.

Any adverse events, including adverse drug reactions, and adverse patient outcomes associated with monitoring tools and patient management will be reported to the Ethics Committee. Should any change to the research protocol required, the Ethics Committee will be informed.

Sample size for each sample is calculated (according to the primary outcomes of the study) as 48 to detect a 20 % difference in time to reach optimal body temperature (expected mean 30 ± 5 minutes, or a 0.3 °C difference in nasopharyngeal temperature when the esophageal temperature reached 37 °C.

In case of missing data (such as due to equipment malfunction, inability to monitor the patient, data not reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results), the participant will be excluded from the study.

The statistical analysis will include descriptive statistics of patient demographics, comparison of both primary outcomes, and comparisons of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled for on-pump coronary artery bypass grafting surgery

Exclusion Criteria:

* Administration of vasopressors during rewarming period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Nasopharyngeal temperature > 37 °C | Rewarming period of cardiopulmonary bypass, usually 30 - 45 minutes
  If the nasopharyngeal temperature is > 37 °C by the time the esophageal temperature reached 37 °C.
Time to 37 °C | Rewarming period of cardiopulmonary bypass, usually 30 - 45 minutes
  Time required to reach an esophageal temperature of 37 °C.

SECONDARY OUTCOMES:
Adverse event: Regional cerebral oxygen saturation | Rewarming period of cardiopulmonary bypass, usually 30 - 45 minutes
  Occurrence and degree of significant drop in regional cerebral oxygen saturation
Length of Intensive Care Unit stay | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from Intensive Care Unit, whichever came first, assessed up to 1 month
  Outcome criteria for coronary artery bypass surgery: length of intensive care unit stay
Length of hospital stay | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 3 months
  Outcome criteria for coronary artery bypass surgery: length of intensive care unit stay
Frequency of atrial fibrillation | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 3 months
  Outcome criteria for coronary artery bypass surgery: occurrence of atrial fibrillation
Frequency of low cardiac output syndrome | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 3 months
  Outcome criteria for coronary artery bypass surgery: occurrence of low cardiac output syndrome
Frequency of stroke | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 3 months
  Outcome criteria for coronary artery bypass surgery: occurrence of stroke
Frequency of delirium | Postoperative period from entrance to Intensive Care Unit until the date of death from any cause or discharge from hospital, whichever came first, assessed up to 3 months
  Outcome criteria for coronary artery bypass surgery: occurrence of postoperative delirium

CONTACTS AND LOCATIONS:
Overall Officials: Başar Erdivanlı, M.D., Principal Investigator — Recep Tayyip Erdogan University Medical Faculty
Locations (1):
- Recep Tayyip Erdogan University, Medical Faculty, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson BW. The hibernator heart--nature's model of resistance to ventricular fibrillation. Cardiovasc Res. 1996 May;31(5):826-32. doi: 10.1016/0008-6363(95)00192-1. PMID 8763414
- [Background] Michenfelder JD, Milde JH. The relationship among canine brain temperature, metabolism, and function during hypothermia. Anesthesiology. 1991 Jul;75(1):130-6. doi: 10.1097/00000542-199107000-00021. PMID 2064037
- [Background] Hori D, Everett AD, Lee JK, Ono M, Brown CH, Shah AS, Mandal K, Price JE, Lester LC, Hogue CW. Rewarming Rate During Cardiopulmonary Bypass Is Associated With Release of Glial Fibrillary Acidic Protein. Ann Thorac Surg. 2015 Oct;100(4):1353-8. doi: 10.1016/j.athoracsur.2015.04.006. Epub 2015 Jul 7. PMID 26163357
- [Background] Engelman R, Hammon JW, Baker RA, Shore-Lesserson L. Rapid Rewarming During Cardiopulmonary Bypass Is Associated With Cerebral Injury. Ann Thorac Surg. 2016 May;101(5):2026-7. doi: 10.1016/j.athoracsur.2015.11.021. No abstract available. PMID 27106452
- [Background] Grigore AM, Grocott HP, Mathew JP, Phillips-Bute B, Stanley TO, Butler A, Landolfo KP, Reves JG, Blumenthal JA, Newman MF; Neurologic Outcome Research Group of the Duke Heart Center. The rewarming rate and increased peak temperature alter neurocognitive outcome after cardiac surgery. Anesth Analg. 2002 Jan;94(1):4-10, table of contents. doi: 10.1097/00000539-200201000-00002. PMID 11772792